CLINICAL TRIAL: NCT04279730
Title: Impact of Fatigue on Physical Performance During a Pulmonary Rehabilitation Program in Patients With COPD
Brief Title: Fatigue and Physical Performance During Pulmonary Rehabilitation
Acronym: PROMOD
Status: Completed | Type: Observational
Sponsor: 5 Santé (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 5S_PROMOD
Record Dates: First submitted 2020-02-12; First posted 2020-02-21 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient pulmonary rehabilitation: Multidisciplinary inpatient pulmonary rehabilitation program lasting 4 weeks (40 sessions, 2 sessions per day, 5 days per week).

SUMMARY:
Patients with COPD benefit from pulmonary rehabilitation (PR), but a ceiling effect of performance (ie. absence of additional exercise tolerance increase) is observed in 80% of patients from only 20 sessions. An imbalance between intensity, duration and frequency of PR sessions, leading to fatigue development in the course of the PR, could explain this ceiling effect. However, previous studies having evaluated the impact of a PR program on fatigue scores reported either a decrease or no changing, but never an increase. To date, no study has evaluated intermediate variations of fatigue score during a PR program, but were limited to a pre-post PR assessment. Therefore, fatigue fluctuations during PR are unknown. Furthermore, most studies had only unidimensional fatigue assessment. Since fatigue is a multifactorial and a multidimensional process, it cannot be accurately estimated through a unique assessment. Given that most of COPD patients do not increase their exercise tolerance from 20 PR sessions, the investigators hypothesize a significant increase of multidimensional fatigue score between the 1st and the 20th PR session during an inpatient rehabilitation program lasting 4 weeks (40 sessions).

DETAILED DESCRIPTION:
Exercise tolerance is an important predictor of health status in patients with chronic obstructive pulmonary disease (COPD). A reduced 6-min walking distance is associated with an increased mortality risk in these patients. Pulmonary rehabilitation (PR) is one of the most efficient strategy to counterac this effect. Patients improving their exercise tolerance after a PR program have a reduced mortality risk. However, exercise tolerance improvement is not systematic after PR, since up to 1/3 of patients do not respond to the intervention. In addition, PR's effects are limited, with a ceiling effect of performance observed in 80% of patients from 20 sessions.

Fatigue could be one candidate to explain the ceiling effect of physical performance during PR. From a theoritical point of view, national and international guidelines on PR have continuously broadened PR interventions for the last 20 years, by progressively introducing in addition to endurance training, resistance training of the lower and then the upper limbs, electrical stimulation, stretching, respiratory muscle training... From a practical point of view, several patients complain of fatigue during PR. However, previous studies having evaluated the impact of a PR program on fatigue scores reported either a decrease or no changing, but never an increase. To date, no study has evaluated intermediate variations of fatigue score during a PR program, but were limited to a pre-post PR assessment. Therefore, fatigue fluctuations during PR are unknown. Furthermore, most studies had only unidimensional fatigue assessment. Since fatigue is a multifactorial and a multidimensional process, it cannot be accurately estimated through a unique assessment. Mutdimensional questionnaires and complementary indicators such as heart rate variability or visuomotor reaction time could be introduced.

Given that most of COPD patients do not increase their exercise tolerance from 20 PR sessions, the investigators hypothesize a significant increase of multidimensional fatigue score between the 1st and the 20th PR session during an inpatient rehabilitation program lasting 4 weeks (40 sessions).

ELIGIBILITY:
Inclusion Criteria:

* Patients admited for a 4-weeks inpatient pulmonary rehabilitation program
* With a confirmed diagnosis of COPD

Exclusion Criteria:

* Severe or unstable heart disease
* Orthopedic, neurologic or psychatric comorbities
* Recent exacerbation (<4 weeks)

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admited for an inpatient PR program at one of the three following pulmonary rehabilitation center will be consecutively recruiting:
  * Clinique du Souffle La Vallonie (Lodève, France)
  * Clinique du Souffle La Solane (Osseja, France)
  * Clinique du Souffle Les Clarines (Riom-es-Montagnes, France)
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Multidimensional fatigue score | Baseline (T0), 1st week (T1), 2nd week (T2), 3rd week (T3) and 4th week (T4) of the PR program
  Change in total fatigue score measured with the MFI-20 questionnaire

SECONDARY OUTCOMES:
6-min walking distance | Baseline (T0), 1st week (T1), 2nd week (T2), 3rd week (T3) and 4th week (T4) of the PR program
  Change in walking distance during a 6-min period over a corridor of 30m length
Heart rate variability | Baseline (T0), 1st week (T1), 2nd week (T2), 3rd week (T3) and 4th week (T4) of the PR program
  Change in SDNN and RMSSD indices of RR intervals during a 5-min resting period and at exercise during a 6-min walking test
Visuomotor reaction time | Baseline (T0), 1st week (T1), 2nd week (T2), 3rd week (T3) and 4th week (T4) of the PR program
  Change in the mean of 15 reaction time in response to visual stimuli
Correlation between fatigue and physical performance | Baseline (T0), 1st week (T1), 2nd week (T2), 3rd week (T3) and 4th week (T4) of the PR program
  Change in the strength of the correlation between indicators of fatigue (muldimensional score, heart rate variability, visuomotor reaction time) and 6-min walking distance

OTHER OUTCOMES:
Physical activity | During the 4 weeks of the PR program (continuous measurement)
  Measurement of physical activity via a triaxial accelerometer
Daily subjective fatigue | Every morning of the 4 weeks PR program
  Fatigue evaluated by the patient every morning with a visual analogic scale

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Heraud, PhD, Study Director — Direction de la recherche et de l'innovation Santé, GCS CIPS, Korian, France
Locations (3):
- France (3):
  - Clinique du Souffle La Vallonie, Lodève
  - Clinique du Souffle La Solane, Osséja
  - Clinique du Souffle Les Clarines, Riom-ès-Montagnes

REFERENCES:
- [Result] Alexandre F, Molinier V, Hognon L, Charbonnel L, Calvat A, Castanyer A, Henry T, Marcenac A, Jollive M, Vernet A, Oliver N, Heraud N. Time-Course of Changes in Multidimensional Fatigue and Functional Exercise Capacity and Their Associations during a Short Inpatient Pulmonary Rehabilitation Program. COPD. 2023 Dec;20(1):55-63. doi: 10.1080/15412555.2022.2164261. PMID 36655947